CLINICAL TRIAL: NCT06751628
Title: Prospective Study of the Methods and Outcomes of CHYME REinstillation After Small Bowel Surgery
Acronym: CHYMERE
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_ED_002
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-07

CONDITIONS: Enterostomy
Keywords: Reinstillation; Small bowel surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Insides system — The miniaturization of the pump proposed by Insides System enables the patient to perform CR independently and to carry the pump anywhere, thus facilitating outpatient implementation of CR.

SUMMARY:
High-output enterocutaneous fistulas (HOF) and double enterostomies are severe complications of abdominal surgery or trauma. Double enterostomies are typically created after small bowel resection in fragile patients who cannot tolerate intestinal reconnection. Reconnection is generally performed 3-6 months later, once patients have regained sufficient healing capacity. In contrast, HOFs occur when intestinal anastomosis healing fails, causing digestive secretions to exit through the abdominal wall. HOFs lead to excessive loss of fluids and nutrients, defined as digestive output exceeding 1500 mL per day for two consecutive days. This often results in severe dehydration and intestinal failure.

Managing HOFs is a complex, resource-intensive process requiring multidisciplinary care to compensate for losses and ensure patient survival. These conditions cause significant patient burden, increase healthcare costs, and often necessitate parenteral nutrition (PN). PN is associated with longer hospital stays, higher risks of central line infections, venous thrombosis, and liver complications (de Vries et al., 2021).

Innovative approaches are needed to restore lost digestive fluids and nutrients in HOF patients. Such solutions could mitigate intestinal failure, reduce PN reliance, prevent dehydration and kidney failure, shorten hospital stays, and improve quality of life by enabling home care. Chyme reinfusion (CR) is an established technique for transferring digestive fluids back into the bypassed intestine (Figure 1A). Historically, this procedure relied on bulky peristaltic pumps available only in specialized centers, with fewer than ten centers in France offering the service. CR has shown significant benefits, with over 85% of patients discontinuing PN and improving nutritional status (Bhat et al., 2020).

A novel, portable pump system developed by Insides System allows patients to independently perform CR and manage their care in outpatient settings. A case series of 10 patients demonstrated that the Insides System enabled PN discontinuation, corrected liver and electrolyte imbalances, and allowed most patients to return home with CR (Sharma et al., 2017).

The CHYMERE study aims to evaluate the effectiveness of chyme reinfusion using a home-compatible device for patients with HOF.

DETAILED DESCRIPTION:
The nutritional data and the quantification of digestive losses will be compared between the period preceding chyme reinfusion (CR) and the CR period using appropriate tests based on the quantitative or qualitative nature of the data. Other endpoints recorded after the start of CR will be analyzed using a descriptive and analytical methodology.

ELIGIBILITY:
Inclusion Criteria:

High-output stoma or enterocutaneous fistula (>1500 mL per day or >1000 mL per day with impact on hydration and nutritional status) Double enterostomy or enterocutaneous fistula with an anatomical configuration allowing chyme reinfusion (CR) Confirmed patency of the downstream digestive segment through digestive contrast imaging

Exclusion Criteria:

Stricture or fistula in the downstream digestive segment Patient refusal to use the device Fine motor or cognitive impairments preventing the patient or a caregiver from handling the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HOF (High-Output Fistulas) who are candidates for chyme reinfusion (CR) using the Insides System device will be included in the study during the pre-implantation consultation or a follow-up consultation. Patient characteristics prior to CR, as well as data related to the objectives mentioned above, will be collected both before device implantation and up to three months after intestinal reconnection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2029-07-14 (Estimated); Study Completion 2030-07-14 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of the Insides System device | 1 year
  reducing the use of parenteral nutrition (median)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided